CLINICAL TRIAL: NCT05408923
Title: Randomized Controlled Trial Comparing Irrisept Versus Normal Saline for Wound Irrigation After Posterior Spine Surgery
Acronym: Irrisept
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It was determined not to be feasible at our site at this time.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Don Moore, MD, PROF, AST CLINICAL DEPT, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2083162
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Spine Degeneration; Cervical Spine Degeneration
MeSH Terms: interventions — Sodium Chloride; chlorhexidine gluconate; Chromogranins

STUDY DESIGN:
Intervention Model Description: Patients will be randomized preoperatively to the study group (Irrisept) versus the control group (sterile saline irrigation).
  Standard betadine and/or chloraprep solution will be used to prep the patient.
  Control group will get normal saline for irrigation throughout the case while study group will be irrigated with the Irrisept solution intermittently throughout the procedure per surgeon discretion.
  No Vancomycin powder will be used in both groups at the time of closure. Standard closure will be performed.
Who Masked: Participant
Masking Description: Irrisept can be differentiated visually from normal saline. Patients will be informed in the consent that they will be blinded to the treatment they are randomized to throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group (Placebo Comparator): Patients in this group will be given the placebo (sterile saline).
  Interventions: Drug: saline 0.9%
- Irrisept (Active Comparator): Patients in this group will be given the study drug (Irrisept).
  Interventions: Drug: (0.05% chlorhexidine gluconate (CHG) in sterile water)

INTERVENTIONS:
Drug: saline 0.9% — Control group will get normal saline for irrigation throughout the case.
  Other Names: sterile saline
  Arms: Placebo Group
Drug: (0.05% chlorhexidine gluconate (CHG) in sterile water) — Intervention group will get Irrisept irrigation (0.05% CHG in sterile water) throughout the case.
  Other Names: Irrisept
  Arms: Irrisept

SUMMARY:
To compare post-operative wound complications in patients randomized to normal saline versus Irrisept solution and any other adverse reactions from the solution.

DETAILED DESCRIPTION:
Wound complications represent a significant risk factor in spinal surgery, particularly in complex multilevel procedures. Surgical site infections (SSI) are the most common health care-associated infection, accounting for 31% of all hospitalized patients with a health care-associated infection. The reported incidence of SSIs following spine surgery ranges from 0.2% to 18.8%. In one study, each episode of wound infection following spine procedure contributed to a mean increase in the cost of care by $4,067 compared to a non-complicated case. The bacteria can adhere to the implants and tissues to create biofilm made by polysaccharide matrix which makes it challenging to clear the infection. Different irrigation techniques and solutions have been utilized to help limit post-operative wound complications. No studies have compared Irrisept solution to normal saline to see if there is a difference in wound complications for posterior spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the University of Missouri hospital system - including the University of Missouri Hospital and Missouri Orthopaedic Institute - with a need for isolated open posterior spine procedures using a posterior open approach.
* Failed conservative treatment - rest, anti-inflammatory medications, physical therapy
* >18 years old and able to provide informed consent

Exclusion Criteria:

* Ongoing or suspected infection
* Revisions of failed back surgeries
* Documented allergy to CHG or CHG products
* Pregnancy - qualitative beta human chorionic gonadotropin (hCG) testing will be performed prior to enrollment
* Prisoners or wards of the state
* Unable to consent to research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Center for Disease Control (CDC)-defined 90-day surgical site infection incidence | 90 days after surgery
  Comparing post-operative surgical site infection incidence between groups for 90 days post-operative using chi-square test.

SECONDARY OUTCOMES:
Wound healing | 90 days after surgery
  Comparing post-operative wound healing incidence between groups for 90 days post-operative using t-Test
Wound complications | 90 days after surgery
  Comparing post-operative wound complications incidence between groups for 90 days post-operative using chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Don Kim Moore, MD, Principal Investigator — University of Missouri - Missouri Orthopaedic Institute
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magill SS, Hellinger W, Cohen J, Kay R, Bailey C, Boland B, Carey D, de Guzman J, Dominguez K, Edwards J, Goraczewski L, Horan T, Miller M, Phelps M, Saltford R, Seibert J, Smith B, Starling P, Viergutz B, Walsh K, Rathore M, Guzman N, Fridkin S. Prevalence of healthcare-associated infections in acute care hospitals in Jacksonville, Florida. Infect Control Hosp Epidemiol. 2012 Mar;33(3):283-91. doi: 10.1086/664048. Epub 2012 Jan 12. PMID 22314066
- [Background] Chahoud J, Kanafani Z, Kanj SS. Surgical site infections following spine surgery: eliminating the controversies in the diagnosis. Front Med (Lausanne). 2014 Mar 24;1:7. doi: 10.3389/fmed.2014.00007. eCollection 2014. PMID 25705620
- [Background] Silber JS, Anderson DG, Vaccaro AR, Anderson PA, McCormick P; NASS. Management of postprocedural discitis. Spine J. 2002 Jul-Aug;2(4):279-87. doi: 10.1016/s1529-9430(02)00203-6. PMID 14589480
- [Background] Rechtine GR, Bono PL, Cahill D, Bolesta MJ, Chrin AM. Postoperative wound infection after instrumentation of thoracic and lumbar fractures. J Orthop Trauma. 2001 Nov;15(8):566-9. doi: 10.1097/00005131-200111000-00006. PMID 11733673
- [Background] Whitmore RG, Stephen J, Stein SC, Campbell PG, Yadla S, Harrop JS, Sharan AD, Maltenfort MG, Ratliff JK. Patient comorbidities and complications after spinal surgery: a societal-based cost analysis. Spine (Phila Pa 1976). 2012 May 20;37(12):1065-71. doi: 10.1097/BRS.0b013e31823da22d. PMID 22045005
- [Background] Onishi Y, Masuda K, Tozawa K, Karita T. Outcomes of an Intraoperative Povidone-Iodine Irrigation Protocol in Spinal Surgery for Surgical Site Infection Prevention. Clin Spine Surg. 2019 Dec;32(10):E449-E452. doi: 10.1097/BSD.0000000000000908. PMID 31609802
- [Background] De Luna V, Mancini F, De Maio F, Bernardi G, Ippolito E, Caterini R. Intraoperative Disinfection by Pulse Irrigation with Povidone-Iodine Solution in Spine Surgery. Adv Orthop. 2017;2017:7218918. doi: 10.1155/2017/7218918. Epub 2017 Oct 2. PMID 29098088
- [Background] Watanabe M, Sakai D, Matsuyama D, Yamamoto Y, Sato M, Mochida J. Risk factors for surgical site infection following spine surgery: efficacy of intraoperative saline irrigation. J Neurosurg Spine. 2010 May;12(5):540-6. doi: 10.3171/2009.11.SPINE09308. PMID 20433302